CLINICAL TRIAL: NCT05097612
Title: "Evaluation of a Soft Exoskeleton With Parallel Springs and Its Ability to Reduce Physical Load During Lifting and Leaning"
Brief Title: Evaluation of a Soft Exoskeleton to Support Forward Leaning and Lifting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Auxivo AG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ETH EK 2021-N-151
Record Dates: First submitted 2021-10-11; First posted 2021-10-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Occupational Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy participant (Experimental): This is a repeated measures design. All participants receive both the intervention and the placebo comparator.
  Interventions: Device: Placebo LiftSuit Exoskeleton; Device: LiftSuit Exoskeleton (low support level); Device: LiftSuit Exoskeleton (medium support level); Device: LiftSuit Exoskeleton (high support level)

INTERVENTIONS:
Device: Placebo LiftSuit Exoskeleton — The LiftSuit is a soft passive wearable device that is designed to support the hip and back muscles during forward leaning and lifting. It exerts it function through Elastic Energy Storages (EES). In this condition the EES are removed from the device to create a placebo device.
Device: LiftSuit Exoskeleton (low support level) — The LiftSuit is a soft passive wearable device that is designed to support the hip and back muscles during forward leaning and lifting. It exerts it function through Elastic Energy Storages (EES). EES of different three different levels of stiffness (low, medium, high stiffness) will be used.
Device: LiftSuit Exoskeleton (medium support level) — The LiftSuit is a soft passive wearable device that is designed to support the hip and back muscles during forward leaning and lifting. It exerts it function through Elastic Energy Storages (EES). EES of different three different levels of stiffness (low, medium, high stiffness) will be used.
Device: LiftSuit Exoskeleton (high support level) — The LiftSuit is a soft passive wearable device that is designed to support the hip and back muscles during forward leaning and lifting. It exerts it function through Elastic Energy Storages (EES). EES of different three different levels of stiffness (low, medium, high stiffness) will be used.

SUMMARY:
In this study the LiftSuit version 2.0 designed by Auxivo AG will be used. The LiftSuit is a soft wearable device that is designed to support workers perform physically demanding tasks including repetitive lifting and working in forward leaning positions. It is put on like a backpack and attached to the body using fabric bands and cuffs. Besides soft fabric parts the LiftSuit contains elastics elements. The elastic elements can be flexibly exchanged by the experimenter. For this experiment elastic elements of known stiffness will be hooked into the fabric frame.

DETAILED DESCRIPTION:
In a first step participants will try on the LiftSuit exoskeleton and adjust it to their body under supervision of the experimenter. When the LiftSuit exoskeleton is adjusted to the participant it is taken off to allow placement of sensors. The sensors used to record heart rate (Polar H9 heart rate monitor, Polar Electro Europe AG, Germany), muscle activity from 8 muscles in the back and hip region (Delsys Trigno, Delsys Europe, United Kingdom) and movement kinematics (OptiTrack motion capture system, NaturalPoint Inc., USA) will be placed by the experimenter (or participant him/herself). To verify that the electromyography sensors, are working and to obtain normalization values, participants will be instructed to conduct maximal voluntary contractions of each muscle that are being recorded. If needed single sensors can be replaced. After this the exoskeleton will be put back on.

ELIGIBILITY:
Inclusion Criteria:

* Included will be volunteers of both sexes within working age (18 to 65 years).

Exclusion Criteria:

* Participants will be excluded if they cannot perform the tasks (squat lifting and forward leaning) due to physical limitations. Furthermore, people who report acute joint or muscle pain or stiffness, or a self-reported history of such problems will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in muscle activity of hip extensor muscles (placebo comparator - low support experimental intervention) | 2 hours
  An elastic band placed external to the body parallel to the spine and over the hip joint is likely to support the muscles that extend the hip and back. Less hip extensor muscle (m. gluteus maximus, hamstrings) activity is expected in LiftSuit conditions compared to the placebo comparator condition.
Change in muscle activity of back extensor muscles (placebo comparator - low support experimental intervention) | 2 hours
  An elastic band placed external to the body paralell to the spine and over the hip joint is likely to support the muscles that extend the hip and back. Less back muscle activity (erector spinae at lumbar and thoracic level) is expected in LiftSuit conditions compared to the placebo comparator condition.

SECONDARY OUTCOMES:
Change in muscle activity of hip extensor muscles related to stiffness level of the Elastic Energy Storages (low, medium, high stiffness). | 2 hours
  A reduction in muscle activity is expected. This reduction is expected to be related to the stiffness level of the EES. With high stiffness, leading to more support, leading to less muscle activity.
Change in muscle activity of back muscles related to stiffness level of the Elastic Energy Storages (low, medium, high stiffness). | 2 hours
  The reduction in muscle activity is expected to be related to the stiffness level of the EES. With high stiffness, leading to more support, leading to less muscle activity.

OTHER OUTCOMES:
Change in muscle activity of abdominal muscles (placebo comparator - experimental intervention) | 2 hours
  An elastic band placed external to the body over the hip joint is likely to support the muscles that extend the hip. It could be that this setup might heightened levels of activity in the abdomen.
Change in hip angle kinematics (placebo comparator - experimental intervention) | 2 hours
  Changed forces around the hip joint might influence movement kinematics of this joint. Changes in position and acceleration of the joint angle will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lambercy, PhD, Principal Investigator — Swiss Federal Institute of Technology
Locations (1):
- ETH Zurich, Rehabilitation Engeineering Laboratory, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Device to be ready for the market